CLINICAL TRIAL: NCT00502723
Title: Prostate Cancer: Multicentric Study Comparing Carcinological and Functional Results of Surgery
Brief Title: Multicentric Study Comparing Carcinological and Functional Results of Surgery
Acronym: PROPENLAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K060402
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2008-01

CONDITIONS: Cancer of the PROSTATE
Keywords: Retropubic Prostatectomy; Surgical Procedures; Laparoscopic
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Radical laparoscopy prostatectomy
  Interventions: Procedure: Radical laparoscopy prostatectomy
- 1 (Experimental): Radical retropubic prostatectomy
  Interventions: Procedure: Radical retropubic prostatectomy

INTERVENTIONS:
Procedure: Radical retropubic prostatectomy — Radical retropubic prostatectomy
  Arms: 1
Procedure: Radical laparoscopy prostatectomy — Radical laparoscopy prostatectomy
  Arms: 2

SUMMARY:
National multicentric prospective open study, comparing two current surgical methods: laparoscopic way versus open retropubic way among patients requiring a radical prostatectomy for a localised prostate cancer.

DETAILED DESCRIPTION:
The aim of this study is to show that radical prostatectomy by laparoscopic way could obtain carcinological results not lower than theses with radical retropubic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male, old patient of less than 70 years,
* having a prostate cancer proven histologically, requiring a radical prostatectomy.
* Clinical stage T1c and rate of PSA (with 20 ng/ml).
* Osseous scintiscanning and abdomen-pelvic scanner negative.
* Patient informed of the study and its participation.
* Patient affiliated to a social security system.

Exclusion Criteria:

* Contra-indication with the surgery or the anaesthesia.
* Antecedent of prostate resection or adenomectomy.
* Antecedent of inguinal hernia treatment.
* Antecedent of deep venous thrombosis of the lower limbs or pulmonary embolism
* Patient privatized of freedom.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
laparoscopic way versus open retropubic way among patients requiring a radical prostatectomy for a localised prostate cancer. | during the study

SECONDARY OUTCOMES:
Carcinological (percentage of positive surgical margins, percentage of capsular crossing). | after the surgical
Functional (urinary continence, sexuality, quality of life) | at 2 years
per and post operational morbidity | during the 36 months
economic | duration and cost of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Claude ABBOU, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Albert Chenevier Henri Mondor, Créteil, France